CLINICAL TRIAL: NCT05931523
Title: Evaluation of the NFFF's Behavioral Health Stress First Aid Intervention
Brief Title: National Fallen Firefighter Foundation's (NFFF) Stress First Aid Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NDRI-USA, Inc. (Other)
Responsible Party: Principal Investigator, Sara Jahnke, Senior Scientist, NDRI-USA, Inc.
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: EMW-2014-FP-00945
Record Dates: First submitted 2023-03-03; First posted 2023-07-05 (Actual); Last update posted 2023-07-10 (Actual); Status verified 2023-07

CONDITIONS: Mental Health Issue

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stress First Aid (Experimental): Fire Departments received the Stress First Aid intervention trainings, tools, and resources.
  Interventions: Behavioral: Stress First Aid
- Wait List Control (No Intervention): Fire Departments in this condition did not receive any intervention or training until the end of their observation year.

INTERVENTIONS:
Behavioral: Stress First Aid — The focus of the model is ongoing monitoring of stress in personnel, wide spread training to help personnel recognize peers or subordinates who may need additional assistance, a spectrum of one-on-one interventions, and the ability to provide personnel higher levels of care when indicated.
  Arms: Stress First Aid

SUMMARY:
Purpose & Aims: Behavioral health interventions implemented to mitigate negative outcomes linked to trauma in the fire service have had limited or iatrogenic effects on firefighters. The National Fallen Firefighters Foundation (NFFF) and the national fire service community have invested considerable resources developing a new behavioral health model to address exposure to traumatic events. The proposed randomized controlled trial will be the first to determine the efficacy of the NFFF's Consensus Protocol on Firefighter Behavioral Health Stress First Aid Intervention (SFAI), as well as evaluating its implementation and acceptability.

Relevance: The SFAI was the result of one of the 16 Firefighter Life Safety Initiatives developed in consultation with the leading fire service organizations in the United States and experts from the traumatic stress research community. Failing to effectively address grief and trauma incidents or symptoms can have devastating effects for firefighters, fire departments, and families. The SFAI was developed to be the national model of trauma intervention to ensure that evidence-based cost-effective care is available to all firefighters.

Methods: Using a cluster randomized clinical trial design (CRCT), experienced scientists and fire service personnel will evaluate the implementation, acceptability, and initial efficacy of the SFAI compared with usual care (i.e., delayed intervention) with 10 fire departments (8 Career, 2 Volunteer) located across the country. Study outcomes include measures assessing implementation of SFAI components, acceptability among firefighters and department leadership, changes in knowledge about and self-efficacy for managing trauma, changes in department morale, and individual firefighter behavioral health outcomes such as symptoms of PTSD and personal growth through coping with traumatic events.

Projected Results & Conclusions: Findings will provide the empirical basis for the newly developed SFAI.

DETAILED DESCRIPTION:
Ten fire departments from across the nation (8 career, 2 volunteer) were recruited for this study. In Aims 1 and 2, program evaluation methods were used to examine the implementation and acceptability of the SFAI intervention components. These evaluation methods were based on standard practices which employs a systematic method for collecting, analyzing, and using information to answer questions about the implementation and acceptability of the SFAI. In Aim 3 a pilot CRCT was conducted comparing the SFAI versus control (delayed treatment) on key behavioral health outcomes. Four career departments were randomized to the SFAI condition and 4 to the control condition. Statistical power analysis was based on these 8 career departments and will provide the primary project outcomes. Between groups outcomes were assessed at 12-months.

ELIGIBILITY:
Inclusion Criteria:

* Firefighters over the age of 18 willing to complete surveys
* Active in a department selected for the study

Exclusion Criteria:

* Those under the age of 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 659 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2018-08 (Actual); Study Completion 2018-10 (Actual)

PRIMARY OUTCOMES:
Acceptability of the SFA training by department personnel using a tailored satisfaction survey | Immediately after training components are delivered and 12 months later
  Percent of trainees who found the training useful and applicable

IPD SHARING:
Plan to Share IPD: Yes
Can be requested from the study team
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: up to 5 years
Access Criteria: Request from research team